CLINICAL TRIAL: NCT02759705
Title: Male Bladder Exstrophy in Adulthood : What Sexuality and Fertility Prospects ?
Brief Title: Bladder Exstrophy (FIVES FertIlity Vesical Exstrophy Sexuality)
Acronym: FIVES
Status: Withdrawn | Type: Observational
Why Stopped: no staff available to do the research
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0044
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Fertility
Keywords: fertility; sexuality; male; exstrophy-epispadias complex; bladder exstrophy; epispadias
MeSH Terms: conditions — Sexuality; Bladder Exstrophy; Epispadias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This analytical descriptive study aims to describe the fertility and sexuality male adult subjects carrying classic bladder exstrophy or epispadias and to highlight infertility risk factors. A questionnaire on paternity, urinary status, erections, ejaculations and sexual self-esteem and a semen analysis will be realized at first consultation, semen analysis results wil be explained at second consultation. It is assumed that fertility and sexuality exstrophic men are impaired.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed the Hospices Civils de Lyon
* Consultant spontaneously in adult or pediatric Urology, or neuroperineal rehabilitation and sexology
* Aged over 18 years
* Born with classic bladder exstrophy or epispadias.

Exclusion Criteria:

* Refusal of participation
* Refusal to sign consent
* minor Patients or protected major, under guardianship
* Patients unable to understand the course of the study
* cloacal exstrophy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male patients born with classic bladder exstrophy or epipadias
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
paternity rate | Baseline (at first consultation)
  paternity rate measured by the ratio of the number of subjects with children to the total number of subjects estimated with questionnaire responses
Sperm quality | up to 2 months
  concentration of mobile live sperm in semen analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Etienne TERRIER, Doctor, Principal Investigator — Urology Department, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, France